CLINICAL TRIAL: NCT07266727
Title: Anesthetic Agent Titration With EEG Wave Analysis: Does it Improve Postoperative Recovery?
Brief Title: Anesthetic Agent Titration With EEG Wave Analysis
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Şeyma Çelik, Principal Investigator, Marmara University
Other Study IDs: 09.2025.25-0113
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Geriatric Patient Care Improvement; EEG Data Analysis
Keywords: electroencephalogram; postoperative delirium; geriatric patients
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Anesthetic Management: Preoperatively, patients were administered the QoR-15 questionnaire and scoring was done according to the Nu-DESC test. Before anesthesia induction, patients will be taught the finger-squeeze test and asked to squeeze the fingers placed in the palm when instructed. If no response is obtained to the test after routine administration of 2 mg/kg propofol and 1.5 mcg/kg fentanyl; 0,5 mg/kg rokuronium administered. Desflurane will be used as maintenance inhalation agent. Hemodynamic parameters and burst suppression time will be recorded at 5-minute intervals during the first 15 minutes after induction and at 15-minute intervals thereafter. At the end of the surgery, the patient will be ready to be sent to the ward with the Modified Aldrete score, and awareness will be assessed with the Modified Brice scale. The QoR-15 questionnaire was repeated at 24 hours postoperatively. For delirium assessment, patients were followed up with the Nu-DESC test for 48 hours postoperatively.
- Anesthetic Management with Kugler EEG method: Preoperatively, patients were administered the QoR-15 questionnaire and scoring was done according to the Nu-DESC test. Before anesthesia induction, patients will be taught the finger-squeeze test and asked to squeeze the fingers placed in the palm when instructed.Patients were administered propofol according to the Kugler EEG analysis (to be kept C-D level) If no response is obtained, fentanyl 1,5 mcg/kg, 0,5 mg/kg rocuronium administered. Desflurane will be used as maintenance inhalation agent. Hemodynamic parameters and burst suppression time will be recorded at 5-minute intervals during the first 15 minutes after induction and at 15-minute intervals thereafter. At the end of the surgery, the patient ready to be sent to the ward with the Modified Aldrete score, and awareness will be assessed with the Modified Brice scale. The QoR-15 questionnaire repeated at 24 hours postoperatively. For delirium assessment, patients followed up with the Nu-DESC test for 48 hours postoperatively.

SUMMARY:
Several studied shown that when general anesthesia is applied under BIS guidance, anesthetic doses are reduced. Additionally it has been found that the risk of postoperative delirium (POD) is reduced and postoperative recovery is accelerated compared to deeper general anesthesia. Current guidelines recommend EEG-based monitoring techniques to prevent postoperative neurocognitive disorders. In clinical practice anesthetic depth is assessed by the patient's autonomic responses to surgical stimulation (pupil diameter, tear, blood pressure and heart rate increase, etc.), the amount of anesthetic gas measured from the expiratory air, and the interpretation of EEG waves and numerical values calculated from these waves (bispactral index, entropy, patient safety index, etc.). The doses of intravenous anesthetic agents used for anesthesia induction are traditionally determined according to body weight. If general anesthetic doses cannot be titrated appropriately for the patients, especially in the elderly and fragile patient group, serious hemodynamic fluctuations may occur during anesthesia induction. The aim of this study is to investigate whether induction and maintenance of anesthesia using the Kugler EEG Analysis method would improve the quality of postoperative recovery in patients aged 65 years and older.

DETAILED DESCRIPTION:
Several studied shown that when general anesthesia is applied under BIS guidance, anesthetic doses are reduced. Additionally it has been found that the risk of postoperative delirium (POD) is reduced and postoperative recovery is accelerated compared to deeper general anesthesia. Current guidelines recommend EEG-based monitoring techniques to prevent postoperative neurocognitive disorders. In clinical practice anesthetic depth is assessed by the patient's autonomic responses to surgical stimulation (pupil diameter, tear, blood pressure and heart rate increase, etc.), the amount of anesthetic gas measured from the expiratory air, and the interpretation of EEG waves and numerical values calculated from these waves (bispactral index, entropy, patient safety index, etc.). The doses of intravenous anesthetic agents used for anesthesia induction are traditionally determined according to body weight. If general anesthetic doses cannot be titrated appropriately for the patients, especially in the elderly and fragile patient group, serious hemodynamic fluctuations may occur during anesthesia induction. The aim of this study is to investigate whether induction and maintenance of anesthesia using the Kugler EEG Analysis method would improve the quality of postoperative recovery in patients aged 65 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and over
* Elective patients undergoing general anesthesia
* EEG monitoring

Exclusion Criteria:

* Pediatric patients
* Patients not giving written consent
* Emergency cases
* History of seizure
* Intracranial surgeries
* Alcohol and substance addiction
* Severe cognitive impairment (dementia, Alzheimer's)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 65 years and older patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Postoperative Recovery Quality | 24 hours
  Data of QoR-15 score in the preoperative period and at the 24th hour postoperatively The 15-item Quality of Recovery (QoR-15) score is a patient-reported outcome measure assessing postoperative recovery. Scores range from 0 to 150, with higher scores indicating better quality of recovery.

SECONDARY OUTCOMES:
Postoperative Delirium Evaluation | 48 hours
  Nu-DESC score in the preoperative period and 48-hour postoperative period The Nursing Delirium Screening Scale (Nu-DESC) is a clinician-rated tool used to screen for delirium. The total score ranges from 0 to 10, with higher scores indicating a worse outcome (greater severity or presence of delirium).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided